CLINICAL TRIAL: NCT06074276
Title: Prospective Randomized Controlled Trial on the Effects of Almond on Facial Skin Collagen and Wrinkles
Brief Title: The Effects of Almond on Facial Skin Collagen and Wrinkles
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Integrative Skin Science and Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: i23-07_Almond_Collagen
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Collagen Degeneration; Wrinkle; Pigmentation; Elastic Skin
MeSH Terms: conditions — Ehlers-Danlos Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Almonds (Experimental): Consumption of almonds 5 times per week
  Interventions: Other: Food: whole almonds
- Control Snack (Placebo Comparator): Consumption of protein and calorie matched non-nut-based food 5 times per week
  Interventions: Other: Food: non-nut snack

INTERVENTIONS:
Other: Food: whole almonds — 60 grams or (~2 oz) will be consumed 5 times per week.
  Arms: Almonds
Other: Food: non-nut snack — Protein and calorie matched non-nut-based food will be consumed 5 times per week by mouth
  Arms: Control Snack

SUMMARY:
Investigate the effects of almond consumption on collagen production, elastin levels, wrinkles, and pigmentation among premenopausal women and postmenopausal women belonging to all Fitzpatrick skin types.

DETAILED DESCRIPTION:
Almonds are energy-dense and rich in beneficial nutrients including B vitamins, vitamin E, mono- and polyunsaturated fatty acids, protein, fiber, minerals and polyphenols. Polyphenols and vitamin E in almonds provide protection to the body in part, through their ability to combat oxidative stress. Clinical studies have demonstrated beneficial effects of almond consumption on diseases such as diabetes and cardiovascular disease.

Almond consumption has been shown to significantly decrease wrinkle severity in two clinical studies conducted with postmenopausal women with Fitzpatrick skin type I and II. Almond intake has also been shown to increase resistance to erythema induced by ultraviolet exposure. The extracellular matrix contains proteins including collagen and elastin, which contributes to the integrity of the skin. Enzymatic and ultraviolet radiation induced degradation and a reduction in synthesis of collagen and elastin contribute to wrinkle formation. Furthermore, the process of menopause decreases the level of estrogen which affects the skin in several ways, including a decrease in skin collagen and hydration, and an increase in wrinkling.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 35 to 70 years of age of all skin types
* 50% of the subjects will be postmenopausal women determined as >1-year loss of menstrual period
* 50% of the subjects will be premenopausal women
* BMI 18.5 - 35 kg/m2
* Individuals with a habitual diet that has been maintained for at least 6 months and to be maintained for the duration of the study
* Individuals must maintain their usual skincare products, defined as products that has been used for at least 1 month, for the duration of the study

Exclusion Criteria:

* Those with a nut allergy
* Those who are unwilling to discontinue oral collagen supplementation 1 month prior to the start of the study
* Individuals who are unwilling to discontinue vitamin E or nut containing supplements 2 weeks prior to and during the intervention.
* Individuals who are pregnant or breastfeeding
* Change in skincare products during the study
* Had a medical or cosmetic procedure such as laser resurfacing or plastic surgery to the face within the last 6 months (include botulinum toxin, dermal fillers, collagen, or other similar cosmetic procedure)
* Has an autoimmune photosensitive condition or known genetic condition with a deficiency in collagen production (such as Ehler-Danlos)
* Those with a skin disease on their face that would affect the assessment of their skin based on the assessment of the investigator.
* Current tobacco smoker or a tobacco smoking history of greater than 10 pack-years

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2023-10-04 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Skin collagen and elastin quantification | 24 weeks
  Assess with biopsy based histological examination
Facial wrinkles | 24 weeks
  Wrinkle severity score measured by Facial Image Analysis System (BTBP 3D image analysis system). Higher scores indicate worsened wrinkle severity and lower scores represent improvement in wrinkle severity.

SECONDARY OUTCOMES:
Pigment intensity score | 12 Weeks
  Change in the appearance of facial pigmentation by high resolution photography (BTBP Clarity Pro) and measures intensity of facial pigmentation. Higher scores indicate darker pigmentation.
Pigment intensity score | 24 Weeks
  Change in the appearance of facial pigmentation by high resolution photography (BTBP Clarity Pro) and measures intensity of facial pigmentation. Higher scores indicate darker pigmentation.
Expression of enzymes that either degrade collagen (MMP1) or inhibit collagen degradation (TIMP1) on skin biopsies | 24 Weeks
  Assess through biopsy based histological examination
Plasma for potential AGE (advanced glycation end products) analysis | 12 Weeks
  Blood samples will be collected
Plasma for potential AGE (advanced glycation end products) analysis | 24 Weeks
  Blood samples will be collected
Facial Wrinkles | 12 Weeks
  Wrinkle severity score measured by Facial Image Analysis System (BTBP 3D image analysis system). Higher scores indicate worsened wrinkle severity and lower scores represent improvement in wrinkle severity.

CONTACTS AND LOCATIONS:
Overall Officials: Raja Sivamani, MD MS AP, Principal Investigator — Integrative Skin Science and Research
Locations (1):
- Integrative Skin Science and Research, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No